CLINICAL TRIAL: NCT03666286
Title: Prospective Registry of Mobilization-, Routine- and Outcome Data of Intensive Care Patients
Acronym: MOBDB
Status: Terminated | Type: Observational
Why Stopped: No further funding to keep up registry.
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Prof. Dr. Stefan Schaller, MD, Senior Specialist Intensive Care, Technical University of Munich
Other Study IDs: MOBDB; DRKS00011576 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2018-09-04; First posted 2018-09-11 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Critical Care; Rehabilitation; Outcome Assessment (Health Care)
Keywords: early mobilization, intensive care, longterm outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intensive Care Patients: Patients >24h on intensive care

SUMMARY:
Registry database of intensive care patients. These data comprises of routine data including mobilization data and follow up assessments.

DETAILED DESCRIPTION:
Registry database of intensive care patients. These data comprises of routine data including mobilization data and follow up assessments.

The database is supposed to help quality improvement as well as

ELIGIBILITY:
Inclusion Criteria:

* Intensive care unit stay > 24 hours

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Intensive Care Unit Patients
Sampling Method: Probability Sample
Enrollment: 1172 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Physical Function at hospital discharge | At hospital discharge, on average within 1 month
  Physical function at ICU discharge with either the mmFIM (minimal modified Functional Independence Measure) or the Barthel subdomains transfer, locomotion and climbing stairs

SECONDARY OUTCOMES:
Hospital Mortality | At hospital discharge, on average within 1 month
  Hospital Mortality
Pre-ICU Function | 2 weeks before ICU admission
  Pre-ICU Function assessed with the WHODAS 2.0 (World Health Organisation's Disability Assessment Schedule), EQ5D (European Quality of Life 5 Dimensions 5 Level) and work details
Global function of the patient | 180 and 360 days after ICU discharge
  Global function of the patient assessed with the WHODAS 2.0 (World Health Organisation's Disability Assessment Schedule)
Physical function of the patient | 180 and 360 days after ICU discharge
  Physical function of the patient assessed with the IADL (The Lawton Instrumental Activities of Daily Living)
Quality of Life of the patient | 180 and 360 days after ICU discharge
  Quality of Life of the patient assessed with the EQ5D (European Quality of Life 5 Dimensions 5 Level)
Cognitive Function | 180 and 360 days after ICU discharge
  Cognitive Function assessed with the MoCA blind (Montreal Cognitive Assessment)
Anxiety and Depression | 180 and 360 days after ICU discharge
  Anxiety and Depression assessed with the IES-R (Impact of Event Scale - Revised) and HADS (Hospital Anxiety and Depression scale)
Return to work | 180 and 360 days after ICU discharge
  Return to work assessed with the WHODAS 2.0 (World Health Organisation's Disability Assessment Schedule)
ICU Mortality | At ICU Discharge, on average within 2 weeks
  ICU Mortality
Physical function at ICU discharge | At ICU Discharge, on average within 2 weeks
  Physical function at ICU discharge with either the mmFIM (minimal modified Functional Independence Measure) or the Barthel subdomains transfer, locomotion and climbing stairs

OTHER OUTCOMES:
Disability-Free survival | 180 and 360 days after ICU discharge
  Disability-Free survival

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Technical University of Munich
Locations (1):
- Klinikum rechts der Isar der TUM, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of anonymous data might be possible on reasonable scientific request.

REFERENCES:
- [Derived] Lorenz M, Fuest K, Ulm B, Grunow JJ, Warner L, Bald A, Arsene V, Verfuss M, Daum N, Blobner M, Schaller SJ. The optimal dose of mobilisation therapy in the ICU: a prospective cohort study. J Intensive Care. 2023 Nov 20;11(1):56. doi: 10.1186/s40560-023-00703-1. PMID 37986100
- [Derived] Fuest KE, Ulm B, Daum N, Lindholz M, Lorenz M, Blobner K, Langer N, Hodgson C, Herridge M, Blobner M, Schaller SJ. Clustering of critically ill patients using an individualized learning approach enables dose optimization of mobilization in the ICU. Crit Care. 2023 Jan 3;27(1):1. doi: 10.1186/s13054-022-04291-8. PMID 36597110